CLINICAL TRIAL: NCT02197052
Title: iScreen Study: Best Methods for Social Screening in Pediatric Caregivers
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: UCSF Benioff Children's Hospital Oakland (Other)
Responsible Party: Sponsor
Other Study IDs: 13-11032
Record Dates: First submitted 2014-07-18; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Disclosure Rates of Social Needs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Computer Based Survey Arm: Participants randomized to the computer based self-completed survey arm were issued a tablet computer to answer survey questions. All participants were encouraged to ask for technical assistance if needed at any point, and like in the face-to-face interviews, electronic survey could be re-initiated at the point of discontinuation after any interruption. Those in the tablet survey arm also could complete the survey in their preferred language and all were additionally given headsets so they could use audio assist with identical, pre-recorded questions in the selected language.
- Face-to-face interview arm: Participants randomized to this condition were interviewed in-person by a fully bilingual (English-Spanish), bi-cultural research assistant trained in cultural humility, standard research protocols and interviewing practices. Interviews were conducted in clinical rooms in respondent's preferred language, were easily interrupted for medical care, and the survey could be re-initiated at the point of discontinuation after any interruption. Participant responses during face-to-face interviews were recorded by the research assistant on paper and later recorded electronically.

SUMMARY:
The goal is to better understand the social needs of a population seeking care in a large, urban children's hospital emergency department with a large Medicaid population. Consenting English and Spanish-speaking adult caregivers will be randomized to social screening via a face -to-face interview with a trained bilingual researcher or via a self-completed tablet-based survey. We hypothesize that there will be no difference in disclosure rates between the two screening formats for items other than highly sensitive items. For highly sensitive items we hypothesize disclosure rates will be higher for the self-completed tablet-based survey.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver must by age 18 years or older accompanying a child less than 18 years old
* Primary language English or Spanish
* Familiar with the child's household environment

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants were drawn from adult caregivers seeking treatment for a child in a fast track arm of a large, urban children's hospital emergency department in Oakland, CA (CHO ED Annex).
Sampling Method: Non-Probability Sample
Enrollment: 552 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Disclosure rates for social needs questions | At time point 1, when the subject is first assessed
  The difference in disclosure rates will be determined by comparing the two arms and determining significant differences for social needs variables.

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Gottlieb, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Children's Hospital Oakland, Oakland, California, United States

REFERENCES:
- [Derived] Gottlieb L, Hessler D, Long D, Amaya A, Adler N. A randomized trial on screening for social determinants of health: the iScreen study. Pediatrics. 2014 Dec;134(6):e1611-8. doi: 10.1542/peds.2014-1439. Epub 2014 Nov 3. PMID 25367545